CLINICAL TRIAL: NCT00047385
Title: National Lung Screening Trial A Randomized Trial Comparing Low-dose Helical CT With Chest Xray for Lung Cancer
Brief Title: National Lung Screening Trial (NLST) Screening
Acronym: NLST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: American College of Radiology Imaging Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NCI-2012-02002; U01CA079778 (NIH); U01CA080098 (NIH); N1CN25476A-85-0-1 (NIH); NIH/NCI (Other: 10 contracts to NCI); CDR0000257938 (Registry Identifier: PDQ [Physician Database Query]); NCT00028808 (obsolete NCT alias)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: small cell lung cancer; non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Tomography, Spiral Computed; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-Dose CT (Experimental)
  Interventions: Device: low-dose helical computed tomography
- Chest X-ray (Experimental)
  Interventions: Device: chest radiography

INTERVENTIONS:
Device: low-dose helical computed tomography — A LDCT is a computerized tomography image with low-dose technique without contrast. The scan is done from the neck to the diaphragm in one breath-hold.
  Other Names: LDCT
  Arms: Low-Dose CT
Device: chest radiography — The chest x-ray in this study was a single posterior-anterior film done with the participant upright.
  Other Names: CXR
  Arms: Chest X-ray

SUMMARY:
RATIONALE: Effective screening tests should help doctors detect lung cancer early and plan curative treatment. It is not yet known whether low-dose helical computed tomography (LDCT) screening is more effective than chest radiography (CXR) screening in reducing death from lung cancer.

PURPOSE: Randomized clinical trial to compare the effectiveness of LDCT scan with that of CXR in screening individuals who are at high risk for developing lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare whether screening with low-dose helical CT scan vs chest x-ray reduces lung cancer-specific mortality in participants who are at high risk for developing lung cancer.

OUTLINE:

NLST participants were randomized to either low-dose helical CT or chest x-ray in equal proportions. A total of 53,454 participants were enrolled (26,722 in low-dose CT and 26,732 in chest radiography) at 33 screening centers across the United States. Screening was offered three times (at baseline and two annual follow-up examinations). The primary endpoint of the study was lung cancer mortality. The study arms were compared with regard to overall mortality, lung cancer incidence, and screening-related complications.

All low-dose scanners and chest x-ray machines were certified for use and met NLST protocol requirements and American College of Radiology guidelines. Low-dose CT acquisitions and chest radiographs were interpreted by trained radiologists. Participants and their health care provider were informed of study examination results. Participants with abnormalities suspicious for lung cancer were contacted for information regarding diagnostic evaluation. Medical records were collected on diagnostic evaluation, medical complications, and initial treatment.

Participants were then contacted at least annually by mail or telephone.

The National Lung Screening Trial (NLST) represents the union of two NCI-sponsored efforts, the NCI Lung Screening Study and the American College of Radiology Imaging Network (ACRIN).

ELIGIBILITY:
Inclusion Criteria:

* Age 55-74 years (pack-years = packs per day * years smoked)
* 30 or more pack-years of cigarette smoking history
* Former smokers: quit smoking within the previous 15 years
* Ability to lie on the back with arms raised over the head
* Signed informed consent form

Exclusion Criteria:

* Metallic implants or devices in the chest or back, such as pacemakers or Harrington fixation rods
* Treatment for, or evidence of, any cancer other than nonmelanoma skin cancer or carcinoma in situ (with the exception of transitional cell carcinoma in situ or bladder carcinoma in situ) in the 5 years prior to eligibility assessment
* History of lung cancer
* History of removal of any portion of the lung, excluding needle biopsy
* Requirement for home oxygen supplementation
* Participation in another cancer screening trial
* Participation in a cancer prevention study, other than a smoking cessation study
* Unexplained weight loss of more than 15 pounds in the 12 months prior to eligibility assessment
* Recent hemoptysis
* Pneumonia or acute respiratory infection treated with antibiotics in the 12 weeks prior to eligibility assessment
* Chest CT examination in the 18 months prior to eligibility assessment

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53454 (Actual)
Dates: Start 2002-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine D. Berg, MD, Study Director — NCI - Early Detection Research Group; Denise R. Aberle, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (33):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Univeristy of California, San Diego, La Jolla, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Pacific Health Research & Education Institute, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Jewish Hopsital Heart and Lung Institute, Louisville, Kentucky
  - Ochsner Medical Foundation Hospital, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota School of Public Health, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Wake Forest University, Winston-Salem, North Carolina
  - St Elizabeth Health Center, Youngstown, Ohio
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Brown University, Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Berg CD, Black WC, Church TR, Fagerstrom RM, Galen B, Gareen IF, Gatsonis C, Goldin J, Gohagan JK, Hillman B, Jaffe C, Kramer BS, Lynch D, Marcus PM, Schnall M, Sullivan DC, Sullivan D, Zylak CJ. The National Lung Screening Trial: overview and study design. Radiology. 2011 Jan;258(1):243-53. doi: 10.1148/radiol.10091808. Epub 2010 Nov 2. PMID 21045183
- [Background] Cody DD, Kim HJ, Cagnon CH, Larke FJ, McNitt-Gray MM, Kruger RL, Flynn MJ, Seibert JA, Judy PF, Wu X. Normalized CT dose index of the CT scanners used in the National Lung Screening Trial. AJR Am J Roentgenol. 2010 Jun;194(6):1539-46. doi: 10.2214/AJR.09.3268. PMID 20489094
- [Background] Clark KW, Gierada DS, Marquez G, Moore SM, Maffitt DR, Moulton JD, Wolfsberger MA, Koppel P, Phillips SR, Prior FW. Collecting 48,000 CT exams for the lung screening study of the National Lung Screening Trial. J Digit Imaging. 2009 Dec;22(6):667-80. doi: 10.1007/s10278-008-9145-9. Epub 2008 Sep 6. PMID 18777192
- [Background] Gierada DS, Garg K, Nath H, Strollo DC, Fagerstrom RM, Ford MB. CT quality assurance in the lung screening study component of the National Lung Screening Trial: implications for multicenter imaging trials. AJR Am J Roentgenol. 2009 Aug;193(2):419-24. doi: 10.2214/AJR.08.1995. PMID 19620438
- [Result] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Result] Singh S, Pinsky P, Fineberg NS, Gierada DS, Garg K, Sun Y, Nath PH. Evaluation of reader variability in the interpretation of follow-up CT scans at lung cancer screening. Radiology. 2011 Apr;259(1):263-70. doi: 10.1148/radiol.10101254. Epub 2011 Jan 19. PMID 21248232
- [Result] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Clapp JD, Clingan KL, Gareen IF, Lynch DA, Marcus PM, Pinsky PF. Baseline characteristics of participants in the randomized national lung screening trial. J Natl Cancer Inst. 2010 Dec 1;102(23):1771-9. doi: 10.1093/jnci/djq434. Epub 2010 Nov 22. PMID 21119104
- [Result] Park ER, Ostroff JS, Rakowski W, Gareen IF, Diefenbach MA, Feibelmann S, Rigotti NA. Risk perceptions among participants undergoing lung cancer screening: baseline results from the National Lung Screening Trial. Ann Behav Med. 2009 Jun;37(3):268-79. doi: 10.1007/s12160-009-9112-9. Epub 2009 Aug 27. PMID 19711141
- [Result] Gierada DS, Pilgram TK, Ford M, Fagerstrom RM, Church TR, Nath H, Garg K, Strollo DC. Lung cancer: interobserver agreement on interpretation of pulmonary findings at low-dose CT screening. Radiology. 2008 Jan;246(1):265-72. doi: 10.1148/radiol.2461062097. Epub 2007 Nov 16. PMID 18024436
- [Derived] Marcinkiewicz AM, Buchwald M, Shanbhag A, Bednarski BP, Killekar A, Miller RJH, Builoff V, Lemley M, Berman DS, Dey D, Slomka PJ. AI for Multistructure Incidental Findings and Mortality Prediction at Chest CT in Lung Cancer Screening. Radiology. 2024 Sep;312(3):e240541. doi: 10.1148/radiol.240541. PMID 39287522
- [Derived] Venkadesh KV, Aleef TA, Scholten ET, Saghir Z, Silva M, Sverzellati N, Pastorino U, van Ginneken B, Prokop M, Jacobs C. Prior CT Improves Deep Learning for Malignancy Risk Estimation of Screening-detected Pulmonary Nodules. Radiology. 2023 Aug;308(2):e223308. doi: 10.1148/radiol.223308. PMID 37526548
- [Derived] Xu K, Khan MS, Li TZ, Gao R, Terry JG, Huo Y, Lasko TA, Carr JJ, Maldonado F, Landman BA, Sandler KL. AI Body Composition in Lung Cancer Screening: Added Value Beyond Lung Cancer Detection. Radiology. 2023 Jul;308(1):e222937. doi: 10.1148/radiol.222937. PMID 37489991
- [Derived] Kinsey CM, Billatos E, Mori V, Tonelli B, Cole BF, Duan F, Marques H, de la Bruere I, Onieva J, San Jose Estepar R, Cleveland A, Idelkope D, Stevenson C, Bates JHT, Aberle D, Spira A, Washko G, San Jose Estepar R. A simple assessment of lung nodule location for reduction in unnecessary invasive procedures. J Thorac Dis. 2021 Jul;13(7):4207-4216. doi: 10.21037/jtd-20-3093. PMID 34422349
- [Derived] Tammemagi MC, Ten Haaf K, Toumazis I, Kong CY, Han SS, Jeon J, Commins J, Riley T, Meza R. Development and Validation of a Multivariable Lung Cancer Risk Prediction Model That Includes Low-Dose Computed Tomography Screening Results: A Secondary Analysis of Data From the National Lung Screening Trial. JAMA Netw Open. 2019 Mar 1;2(3):e190204. doi: 10.1001/jamanetworkopen.2019.0204. PMID 30821827
- [Derived] Wong JYY, Bassig BA, Seow WJ, Hu W, Ji BT, Blair A, Silverman DT, Lan Q. Lung cancer risk in welders and foundry workers with a history of heavy smoking in the USA: The National Lung Screening Trial. Occup Environ Med. 2017 Jun;74(6):440-448. doi: 10.1136/oemed-2016-104168. Epub 2017 Jan 9. PMID 28069970
- [Derived] Patz EF Jr, Greco E, Gatsonis C, Pinsky P, Kramer BS, Aberle DR. Lung cancer incidence and mortality in National Lung Screening Trial participants who underwent low-dose CT prevalence screening: a retrospective cohort analysis of a randomised, multicentre, diagnostic screening trial. Lancet Oncol. 2016 May;17(5):590-9. doi: 10.1016/S1470-2045(15)00621-X. Epub 2016 Mar 18. PMID 27009070
- [Derived] Marcus PM, Doria-Rose VP, Gareen IF, Brewer B, Clingan K, Keating K, Rosenbaum J, Rozjabek HM, Rathmell J, Sicks J, Miller AB. Did death certificates and a death review process agree on lung cancer cause of death in the National Lung Screening Trial? Clin Trials. 2016 Aug;13(4):434-8. doi: 10.1177/1740774516638345. Epub 2016 Mar 22. PMID 27006427
- [Derived] Tanner NT, Gebregziabher M, Hughes Halbert C, Payne E, Egede LE, Silvestri GA. Racial Differences in Outcomes within the National Lung Screening Trial. Implications for Widespread Implementation. Am J Respir Crit Care Med. 2015 Jul 15;192(2):200-8. doi: 10.1164/rccm.201502-0259OC. PMID 25928649
- [Derived] Clark MA, Gorelick JJ, Sicks JD, Park ER, Graham AL, Abrams DB, Gareen IF. The Relations Between False Positive and Negative Screens and Smoking Cessation and Relapse in the National Lung Screening Trial: Implications for Public Health. Nicotine Tob Res. 2016 Jan;18(1):17-24. doi: 10.1093/ntr/ntv037. Epub 2015 Mar 6. PMID 25746779
- [Derived] Black WC. Computed tomography screening for lung cancer in the National Lung Screening Trial: a cost-effectiveness analysis. J Thorac Imaging. 2015 Mar;30(2):79-87. doi: 10.1097/RTI.0000000000000136. PMID 25635704
- [Derived] Black WC, Gareen IF, Soneji SS, Sicks JD, Keeler EB, Aberle DR, Naeim A, Church TR, Silvestri GA, Gorelick J, Gatsonis C; National Lung Screening Trial Research Team. Cost-effectiveness of CT screening in the National Lung Screening Trial. N Engl J Med. 2014 Nov 6;371(19):1793-802. doi: 10.1056/NEJMoa1312547. PMID 25372087
- [Derived] Osinusi A, Kohli A, Marti MM, Nelson A, Zhang X, Meissner EG, Silk R, Townsend K, Pang PS, Subramanian GM, McHutchison JG, Fauci AS, Masur H, Kottilil S. Re-treatment of chronic hepatitis C virus genotype 1 infection after relapse: an open-label pilot study. Ann Intern Med. 2014 Nov 4;161(9):634-8. doi: 10.7326/M14-1211. PMID 25364884
- [Derived] Pinsky PF, Gierada DS, Hocking W, Patz EF Jr, Kramer BS. National Lung Screening Trial findings by age: Medicare-eligible versus under-65 population. Ann Intern Med. 2014 Nov 4;161(9):627-33. doi: 10.7326/M14-1484. PMID 25199624
- [Derived] Aberle DR, DeMello S, Berg CD, Black WC, Brewer B, Church TR, Clingan KL, Duan F, Fagerstrom RM, Gareen IF, Gatsonis CA, Gierada DS, Jain A, Jones GC, Mahon I, Marcus PM, Rathmell JM, Sicks J; National Lung Screening Trial Research Team. Results of the two incidence screenings in the National Lung Screening Trial. N Engl J Med. 2013 Sep 5;369(10):920-31. doi: 10.1056/NEJMoa1208962. PMID 24004119
- [Derived] National Lung Screening Trial Research Team; Church TR, Black WC, Aberle DR, Berg CD, Clingan KL, Duan F, Fagerstrom RM, Gareen IF, Gierada DS, Jones GC, Mahon I, Marcus PM, Sicks JD, Jain A, Baum S. Results of initial low-dose computed tomographic screening for lung cancer. N Engl J Med. 2013 May 23;368(21):1980-91. doi: 10.1056/NEJMoa1209120. PMID 23697514
- [Derived] Singh SP, Gierada DS, Pinsky P, Sanders C, Fineberg N, Sun Y, Lynch D, Nath H. Reader variability in identifying pulmonary nodules on chest radiographs from the national lung screening trial. J Thorac Imaging. 2012 Jul;27(4):249-54. doi: 10.1097/RTI.0b013e318256951e. PMID 22627615
- [Derived] Matsuoka S, Washko GR, Dransfield MT, Yamashiro T, San Jose Estepar R, Diaz A, Silverman EK, Patz S, Hatabu H. Quantitative CT measurement of cross-sectional area of small pulmonary vessel in COPD: correlations with emphysema and airflow limitation. Acad Radiol. 2010 Jan;17(1):93-9. doi: 10.1016/j.acra.2009.07.022. Epub 2009 Sep 30. PMID 19796970
- [Derived] Dransfield MT, Washko GR, Foreman MG, Estepar RS, Reilly J, Bailey WC. Gender differences in the severity of CT emphysema in COPD. Chest. 2007 Aug;132(2):464-70. doi: 10.1378/chest.07-0863. Epub 2007 Jun 15. PMID 17573503
- See also: Web site for additional information — http://www.cancer.gov/nlst

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from August 2002 through April 2004 at 33 NLST sites.
Pre-assignment Details: Participants signed a study informed consent prior to being randomized to a study arm.
Groups:
- Low-Dose CT: Participants undergo low-dose helical CT examination.
- Chest X-ray: Participants undergo chest x-ray examination.
Period: Overall Study
Arm/Group | Low-Dose CT | Chest X-ray
Started | 26722 | 26732
Completed | 26455 (Had at least one screening exam.) | 26232
Not Completed | 267 | 500
Not completed — Death before any screening | 2 | 5
Not completed — Lung Cancer diagnosed before screening | 5 | 3
Not completed — Eligible for screening but had no screen | 260 | 492

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose CT | Chest X-ray | Total
Number analyzed (Participants) | 26722 | 26732 | 53454
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19612 | 19622 | 39234
  >=65 years | 7110 | 7110 | 14220
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (5.0) | 61.4 (5.0) | 61.4 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10952 | 10970 | 21922
  Male | 15770 | 15762 | 31532
Region of Enrollment [Number; unit: participants]
  United States | 26,722 | 26,732 | 53454

OUTCOME MEASURES:

1. Primary Outcome: Lung Cancer Deaths
Description: Lung cancer deaths confirmed in participants by Endpoint Verification if available, otherwise by death certificate.
Time Frame: All events through December 31, 2009; median follow-up 6.5 years.
Population: All participants randomized were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Groups:
- LDCT Screening: Participants randomized to receive three annual low-dose helical CT exams of the chest.
- CXR Screening: Participants randomized to receive three annual chest radiographs.
Arm/Group | LDCT Screening | CXR Screening
Number analyzed (Participants) | 26722 | 26732
Participants | 356 | 443
Statistical Analysis 1: Comparison: LDCT Screening vs CXR Screening; Alternative hypothesis: LDCT screening reduces lung cancer mortality relative to chest x-ray. Power: 90% for a 20% reduction in lung cancer mortality; Test type: Superiority or Other; p = 0.004, Weighted log-rank (details below) — P-value is adjusted for multiple comparisons; Weights in weighted log-rank statistic increased linearly from zero at randomization to full weight at 4 years and thereafter; Hazard Ratio (HR) = 0.800, 95% CI 2-sided [0.733 to 0.932]

2. Secondary Outcome: Deaths From All Causes in All Randomized Participants.
Description: Deaths from all causes were compared between the low-dose CT group and the chest radiography group among all randomized participants.
Time Frame: All events through December 31, 2009; median follow-up 6.5 years.
Population: All participants randomized were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | LDCT Screening | CXR Screening
Number analyzed (Participants) | 26722 | 26732
Participants | 1877 | 2000
Statistical Analysis 1: Comparison: LDCT Screening vs CXR Screening; Alternative hypothesis: LDCT screening reduced all-cause mortality relative to chest x-ray; Test type: Superiority or Other; p = 0.02, Weighted log-rank (details below) — No adjustment for multiple comparisons. Only one analysis performed; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.933, 95% CI 2-sided [0.864 to 0.988]

3. Secondary Outcome: Lung Cancer Diagnoses
Description: Lung cancer diagnoses confirmed by medical record abstraction.
Time Frame: All events through December 31, 2009; median follow-up 6.5 years
Population: All participants randomized were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | LDCT Screening | CXR Screening
Number analyzed (Participants) | 26722 | 26732
Participants | 1060 | 941
Statistical Analysis 1: Comparison: LDCT Screening vs CXR Screening; Test type: Superiority or Other; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [1.03 to 1.23] — Denominator: LDCT Group Numerator: CXR Group

4. Secondary Outcome: Complications of Diagnostic Evaluation Following a Positive Screening Test.
Description: Number of participants who experienced complications during diagnostic work-up of a screening CT or CXR that was suspicious for lung cancer.
Time Frame: One year from screening examination
Population: The units analyzed were positive screening exams with documented diagnostic follow-up. If participant received 3 positive screens with documented follow-up after each one, he/she would be counted 3 times in the number of units analyzed.
Measure: Number; unit: Pos. screens w/ complications
Units Other Than Participants: Positive Screens with Follow-up
Arm/Group | LDCT Screening | CXR Screening
Number analyzed (Participants) | 26722 | 26732
Number analyzed (Positive Screens with Follow-up) | 17702 | 4953
Pos. screens w/ complications | 245 | 81

5. Secondary Outcome: T0 (Baseline) Screening Results
Description: Results of radiologist's interpretation of images from LDCT or CXR screening exam at T0.
Time Frame: T0 (at study entry)
Population: All participants randomized were analyzed.
Measure: Number; unit: Participants
Arm/Group | LDCT Screening | CXR Screening
Number analyzed (Participants) | 26722 | 26732
Participants
  Positive | 7191 | 2387
  Significant abnor. not suspicious for lung cancer | 2695 | 785
  No, or minor abnormality | 16423 | 22863
  Eligible but not screened | 406 | 689
  Not eligible for screen | 7 | 8

6. Secondary Outcome: T1 Screening Results
Description: Results of radiologist's interpretation of images from LDCT or CXR screening exam at T1. Includes a comparison with images from T0 screen.
Time Frame: T1 (one year after entry)
Population: All participants randomized were analyzed
Measure: Number; unit: Participants
Arm/Group | LDCT Screening | CXR Screening
Number analyzed (Participants) | 26722 | 26732
Participants
  Positive | 6901 | 1482
  Significant abnor. not suspicious for lung cancer | 1519 | 429
  No, or minor abnormality | 16295 | 22178
  Eligible but not screened | 1570 | 2321
  Not eligible for screen | 437 | 322

7. Secondary Outcome: T2 Screening Results
Description: Results of radiologist's interpretation of images from LDCT or CXR screening exam at T2. Includes a comparison with images from T0 and T1 screens.
Time Frame: T2 (two years after entry)
Population: All participants randomized were analyzed
Measure: Number; unit: Participants
Arm/Group | LDCT Screening | CXR Screening
Number analyzed (Participants) | 26722 | 26732
Participants
  Positive | 4054 | 1174
  Significant abnor. not suspicious for lung cancer | 1408 | 361
  No, or minor abnormality | 18640 | 21811
  Eligible but not screened | 1840 | 2764
  Not eligible for screen | 780 | 622

ADVERSE EVENTS:
Time Frame: During each annual screening visit.
Description: These events are solely those prompted by the screening examination.
Arm/Group | Low-Dose CT | Chest X-ray
Serious Adverse Events (participants affected / at risk) | 0/26722 | 2/26732
Other Adverse Events (participants affected / at risk) | 0/26722 | 0/26732
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose CT (N=26722) | Chest X-ray (N=26732)
Nausea/vomiting, bradycardia, diaphoresis (General disorders) | 0 (0) | 1 (1) — Transient syncope w/ vomiting/bradycardia/diaphoresis/ashen color after phlebotomy and single forced expiration for spirometry. Hospitalized for monitoring; MI ruled out. Recovered with time, rest, and liquids.
Cardiac symptoms (Cardiac disorders) | 0 (0) | 1 (1) — Shortness of breath, diaphoresis, jaw pain and general cardiac symptoms. Admitted to hospital; MI ruled out. Treated with medication/inhalers for COPD exacerbation. Stable through the admission; fully recovered the following day.

LIMITATIONS AND CAVEATS:
NLST utilized institutions with special expertise. The "healthy volunteer" effect may apply. Scanners are now more technologically advanced. Ongoing LDCT screening may reduce the rate of lung cancer deaths more than three rounds done in NLST.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less